CLINICAL TRIAL: NCT07016581
Title: Optimal Duration of Spinal Cord Stimulation Trial Procedure: Length and Diagnostic Accuracy
Status: Enrolling by invitation | Type: Observational
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: Mayo Clinic (Other); Ohio State University (Other); M.D. Anderson Cancer Center (Other)
Responsible Party: Principal Investigator, Jay Karri, Principal Investigator, University of Maryland, Baltimore
Other Study IDs: HP-00113001
Record Dates: First submitted 2025-06-04; First posted 2025-06-11 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Chronic Pain
Keywords: spinal cord stimulation; spinal cord stimulation trial
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study Cohort: Adult patients with chronic pain undergoing an spinal cord stimulation trial procedure
  Interventions: Diagnostic Test: Daily survey

INTERVENTIONS:
Diagnostic Test: Daily survey — All patients undergoing an spinal cord stimulation trial procedure (which will be conducted in accordance to standard clinical practices per site) will be given daily surveys to assess their analgesic and functional benefit.

SUMMARY:
This study aims to find out the optimal duration (in days) needed for a spinal cord stimulator (SCS) trial procedure for treating chronic pain. While shorter trial periods could lower risks like infections or bleeding (especially for patients who need to stop blood thinners), patients also need sufficient time to achieve meaningful pain and function relief, and to report willingness to proceed to permanent implantation. Unfortunately, the optimal duration of an SCS trial procedure is not currently known. We aim to explore this optimal duration across a multi-center study by studying daily surveys completed across the duration of SCS trial procedures.

DETAILED DESCRIPTION:
Spinal cord stimulation (SCS) is a well-established therapy for chronic pain. However before one can proceed with SCS as a permanent therapy, they must undergo an antecedent SCS trial procedure to assess its effectiveness as a treatment for the patient's pain. The SCS trial procedure involves the percutaneous placement of leads with electrical contacts into the epidural space.

Given the infectious risks associated with an SCS trial, including those associated with significant morbidity and mortality, the typical duration of an SCS trial procedure ranges from 3 to 14 days. Additionally, given the risks for epidural hematoma formation, patients on certain anti-platelet and anti-coagulant medications require medication cessation prior to and across the SCS trial duration. In these scenarios, prolonging the withholding of these medications can place these patients at serious risks for serious embolic and/or vascular events. However, while reducing the duration an SCS trial procedure may help mitigate the risks for serious infectious and embolic and/or vascular events, patients with chronic pain conditions may typically need several days to achieve and report meaningful analgesic and functional responses and willingness to proceed with a permanent SCS implantation procedure. However, the optimal duration required for an SCS trial response has yet to be clearly established.

In this study, we aim to explore the optimal duration of the SCS trial procedure and assess how daily pain levels and patient satisfaction impact the decision to permanently implant a SCS device. The primary objective is to determine the optimal number of days required to accurately predict SCS trial procedure outcomes.

This prospective, multi-center study will enroll a target of 100 patients undergoing an SCS trial procedure (conducted in accordance to standard clinical practices per site). In addition to demographics, Patient-Reported Outcomes Measurement Information System (PROMIS) scores, SCS e-health tool recommendations, and key SCS parameters, patients will complete daily surveys to assess their analgesic and functional benefit across the duration of the SCS trial. Analyses will be performed to determine: 1) the number of days it takes to define final trial outcomes (for positive responders and not-positive responders); 2) if and how PROMIS domains correlate with days to define final trial outcomes; and 3) if and how SCS e-health tool recommendations correlate with days to define final trial outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years old, with capacity for study consent
* Clinical evidence of a chronic pain condition amenable for treatment with spinal cord stimulation
* Chronic pain duration >12 weeks

Exclusion Criteria:

* Pregnancy
* Worker's compensation status
* Previously failed spinal cord stimulation trial
* Chronic opioid use with >50 morphine milligram equivalents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with chronic pain undergoing an spinal cord stimulation trial procedure to assess for candidacy for permanent implantation of an spinal cord stimulation device.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-06-05 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Days to Achieve Response to Spinal Cord Stimulation Trial Procedure | 3-14 days
  minimum number of days required to accurately predict spinal cord stimulation trial outcomes (positive or negative)

CONTACTS AND LOCATIONS:
Overall Officials: Jay Karri, MD, MPH, Principal Investigator — University of Maryland; Ryan D'Souza, MD, Principal Investigator — Mayo Clinic
Locations (4):
- United States (4):
  - University of Maryland, Baltimore, Maryland
  - Mayo Clinic, Rochester, Minnesota
  - Ohio State University, Columbus, Ohio
  - MD Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: Undecided